CLINICAL TRIAL: NCT01244997
Title: Prospective Evaluation of Immediate Temporized Implants
Brief Title: Evaluation of Implants Placed Immediately or Delayed Into Extraction Sites
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Michael S. Block DMD, LSU School of Dentistry
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB4729
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2010-11

CONDITIONS: Dental Caries
Keywords: Partial edentulism; Bone atrophy; Bone healing
MeSH Terms: conditions — Dental Caries | interventions — Dental Implants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate implant placement (Experimental): This arm is an immediate placement of a dental implant following tooth extraction.
  Interventions: Procedure: Dental Implant
- Delayed Implant (Active Comparator): This is the traditional method for implants. This arm will be done following a healing of the area.
  Interventions: Procedure: Dental Implant

INTERVENTIONS:
Procedure: Dental Implant — This is designed to compare the response of the crestal bone after implants are placed whether delayed or immediately after tooth extraction in the maxilla.

SUMMARY:
IRB4729 Study Hypothesis: Is there a significant difference in the hard and soft tissue response comparing immediate with delayed implant after tooth removal, with immediate provisionalization, in maxillary anterior sites.

The purpose of this study is to determine and compare the crestal bone levels as the primary endpoint variable for implants placed and temporized in extraction sites, to implants placed into extraction sites after the extraction site has been grafted and healed for 4 months, all immediately restored with an anatomic provisional restoration.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be willing to be present for examination two times a year for at least three years, as well as maintenance cleaning twice a year 3 months prior to the data collection visit
* All patients will be free of uncontrolled diabetes (any type, existing malignancy, and will not be receiving any therapy that suppresses their immune system, such as radiation, chemotherapy, or chronic steroid usage
* Need for extraction of a single rooted maxillary central or lateral incisor, canine, or premolar, with no signs of acute infection (purulent exudate, erythema, pain and swelling).
* Patients will have bone present on all surfaces of the tooth within 3mm of the gingival margin of the planned restoration, in order to provide sufficient bone to circumferentially cover the implant.
* all patients will have adequate space for satisfactory restoration of the edentulous space.
* each patients dentition will be free of active periodontal disease or exhibit controllable periodontal disease such that their teeth will clinically be non-mobile and have probing depths less than 3mm.
* All prospective sites will have at least 2mm of attached or keratinized gingiva.
* The crestal bone width should be enough to accommodate either a 3.75mm diameter implant for the central incisor, canine, and premolar sites or a 3.25 mm diameter implant for the lateral incisor tooth sites. Bone heights should be at least 14mm for accommodation of the implant.

Exclusion Criteria:

* Patients with labial dehiscence defects greater than 3mm from the proposed gingival margin of the planned restoration will be excluded from this study.
* Patients who cannot come for follow up due to conflicts of schedules will not be accepted into the study.
* Patients with advanced cardiovascular, pulmonary, renal, liver disease that place them in an ASA III or IV rating will be excluded. Post-menopausal women with known osteoporosis as determined by their medical internist, will be excluded. Patients with known alcohol abuse will be excluded.

Ages: 21 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2003-11; Primary Completion 2008-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Crestal bone levels adjacent to the implants | 24 months
  An evaluation of crestal bone level changes when implants are placed into extraction sites. Levels will be measured on standardized digital radiographs of the implants using their threads as a monitor of magnification and a preextraction reference in the measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- LSU School of Dentistry, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Ryser MR, Block MS, Mercante DE. Correlation of papilla to crestal bone levels around single tooth implants in immediate or delayed crown protocols. J Oral Maxillofac Surg. 2005 Aug;63(8):1184-95. doi: 10.1016/j.joms.2005.04.025. PMID 16094589